CLINICAL TRIAL: NCT07163793
Title: A Pilot Study of Reduced Venetoclax Exposure in Patients With Acute Myeloid Leukemia in Complete Remission
Brief Title: Pilot Study of Reduced Venetoclax Exposure
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-0579
Record Dates: First submitted 2025-08-07; First posted 2025-09-09 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Acute Myeloid Leukemia in Remission
Keywords: AML
MeSH Terms: interventions — Azacitidine; Decitabine; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Azacytadine + Venetoclax (Active Comparator)
  Interventions: Drug: Azacitidine; Drug: Venetoclax
- Decitabine + Venetoclax (Active Comparator)
  Interventions: Drug: Decitabine; Drug: Venetoclax

INTERVENTIONS:
Drug: Azacitidine — Given Day 1-7 with Venetoclax Day 1-14 every 28 days until off study
  Other Names: Vidaza
  Arms: Azacytadine + Venetoclax
Drug: Decitabine — Given Day 1-5 with Venetoclax Day 1-14 every 28 days until off
  Other Names: Dacogen
  Arms: Decitabine + Venetoclax
Drug: Venetoclax — Venetoclax up to 400mg a day on Day 1-14 every 28 days until off in combination with Azacitidine or Decitabine
  Other Names: Venclexta, Venclyxto

SUMMARY:
Pilot Study of Reduced Venetoclax Exposure

DETAILED DESCRIPTION:
A pilot single-arm clinical trial is proposed to assess the primary objective: the tolerability of 14-day Venetoclax cycles in acute myeloid leukemia (AML) patients who have achieved remission and are ineligible for intensive treatment. Participants in the study will transition to a maintenance regimen that reduces the Venetoclax dosage to 14 days per cycle while continuing the hypomethylating agent (HMA) used during induction. Treatment cycles will occur every 28 days. Participants will continue treatment on study until experiencing a grade 4 cytopenic event lasting more than 7 days, an adverse event requiring regimen modification, relapse, or death.

Our primary hypothesis posits that AML patients receiving Venetoclax for 14 days per cycle will exhibit improved treatment tolerability with a reduced rate of grade 4 cytopenia compared to historical data from the VIALE A trial.

ELIGIBILITY:
Inclusion Criteria:

1. Stated willingness to comply with all study procedures and availability for the duration of the study
2. Ability to take oral medication and be willing to adhere to the study regimen
3. Diagnosed by current WHO or ICC criteria with Acute Myeloid Leukemia and treated for initial induction therapy with one of two regimens:

   1. 5-Azacitidine administered subcutaneously at a dose of 75mg/m2/day X 7 days in combination with VEN (21-28 days/cycle)
   2. Decitabine administered intravenously at a dose of 20mg/m2/day administered in combination with VEN (21-28 days/cycle)
4. Achieving morphological CR/CRi by bone marrow biopsy with <5% blasts within 3 cycles. See Appendix 2 for definitions.
5. Consent to be obtained within 10 days (+/- 3 days) of bone marrow biopsy report showing morphological remission. C1D1 of trial to be initiated within 10 days (+/- 7 days) of bone marrow biopsy report showing morphological remission.
6. ECOG 0-3
7. Intensive treatment ineligible; transplant ineligible or refusal of transplant
8. Patient must be able to understand and sign informed consent and additional study documents
9. On C1D1 of trial, patient must have count recovery with ANC >1000, platelets > 50, Hemoglobin > 7.7 and without transfusion support for 7 days.
10. No growth factor (G-CSF) use in 14 days prior to C1 D1 of trial.

Exclusion Criteria:

1. Treatment with another investigational drug
2. Use of growth factor (G-CSF) within the last 14 days prior to C1D1 of trial treatment.
3. On concomitant targeted therapy such as FLT3 inhibitor or IDH1/2 inhibitor.
4. Subject has received treatment prior to induction with the following:

   i. Prior hypomethylating agent or BCL-2 inhibitor for either AML or MDS other than for induction prior to enrollment.

   ii. Prior CAR-T cell therapy. iii. Experimental or investigational drug therapy for 14 days prior to study entry leukemia-directed therapies.
5. Subject has:

   i. Acute promyelocytic leukemia (APL) with t(15;17). ii. Presence of t(9;22) given the potential indication for concurrent tyrosine kinase therapy.

   iii. Known active CNS involvement with AML.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-10-07 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Venetoclax Tolerability Rate | 12 months
  Tolerability rate defined as the proportion of patients who do not experience grade 4 neutropenia (per the CTCAE v5.0) for over 7 continuous days within the first three cycles of maintenance therapy (90 days).
  Patient will be evaluated on Day 1 of each cycle. Laboratory studies of prior cycle will be reviewed on that day to identify if patient had >7 continuous days of cytopenia.

SECONDARY OUTCOMES:
Evaluation of Event-Free Survival (EFS) | 12 months
  EFS: Time from treatment-to-treatment discontinuation, relapse, death of any cause, or lost to follow up (Lost to follow up defined as missing scheduled appointment with no response to 3 phone calls and 1 certified letter).
Time to Detriment | 48 months
  Time to detriment defined as time to meaningful change in the EORTC-QLQ-C30. A meaningful change is defined as a decrease by at least 10 points from their baseline evaluation
  The EORTC-QLQ0-C30 will be filled out by patient on Day 1 of every cycle for the first 12 cycles of maintenance therapy.
Number of pRBC transfusion | 48 months
  Number of pRBC transfusion received while on trial therapy.
  Number of platelet transfusion received while on trial therapy.
  Number of transfusions to be described per patient year.
  Data collected on Day 1 of every cycle.
Evaluate Number of Hospital Admissions | 12 months
  To be evaluated at time of trial therapy discontinuation or 12 cycles of therapy, whichever occurs first.
Rate of adverse events/toxicities | 48 months
  dverse events/Toxicities related to treatment.
  List of adverse events/toxicities expected listed in Section 8.
Evaluation of Relapse-Free Survival (RFS) | 12 months
  RFS: Time from treatment initiation to relapse, death, or lost to follow up (Lost to follow up defined as missing scheduled appointment with no response to 3 phone calls and 1 certified letter).
Evaluation of Overall Survival (OS) | 12 months
  OS: Time to death or lost to follow up (Lost to follow up defined as missing scheduled appointment with no response to 3 phone calls and 1 certified letter)
Evaluate Number of Days Admitted | 12 months
  To be evaluated at time of trial therapy discontinuation or 12 cycles of therapy, whichever occurs first.
Evaluate Number of Unanticipated lab appointments | 12 months
  To be evaluated at time of trial therapy discontinuation or 12 cycles of therapy, whichever occurs first.
Evaluate Number of Unanticipated clinic visits | 12 months
  To be evaluated at time of trial therapy discontinuation or 12 cycles of therapy, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Boiclair Stephanie, MD, Principal Investigator — Northwell Health
Locations (1):
- Zuckerberg Cancer Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No